CLINICAL TRIAL: NCT01260610
Title: An Exploratory, Randomized, Controlled Study of Tenofovir Plus Telbivudine Versus Monotherapy With Either Drug Alone in HBeAg Negative Chronic Hepatitis B Patients
Brief Title: Randomized Controlled Study of Tenofovir Plus Telbivudine Versus Monotherapy With Either Drug in HBeAg Negative Chronic Hepatitis B Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of funds
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLDT600AIN05T
Record Dates: First submitted 2010-12-14; First posted 2010-12-15 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2011-06

CONDITIONS: Chronic Hepatitis B
Keywords: Hepatitis B, Tenofovir, Telbivudine
MeSH Terms: conditions — Hepatitis B, Chronic; Hepatitis B | interventions — Tenofovir; Telbivudine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tenofovir (Active Comparator)
  Interventions: Drug: Tenofovir
- Telbivudine (Active Comparator)
  Interventions: Drug: Telbivudine
- Tenofovir plus Telbivudine (Experimental)
  Interventions: Drug: Tenofovir plus Telbivudine

INTERVENTIONS:
Drug: Tenofovir — 300 mg of Tenofovir daily
  Arms: Tenofovir
Drug: Telbivudine — 600 mg of Telbivudine daily
  Arms: Telbivudine
Drug: Tenofovir plus Telbivudine — Tenofovir (300 mg daily) plus Telbivudine (600 mg daily)
  Arms: Tenofovir plus Telbivudine

SUMMARY:
Combination therapies using nucleos(t)ide analogues lead to higher viral suppression although it may not be sustained for long. Also it remains unknown if combination of more potent analogues is more beneficial than individual drugs. Thus this study is carried out to determine the efficacy and safety of combination of tenofovir plus telbivudine (two most potent nucleos(t)ide analogues)versus monotherapy with either drug alone. This is a 104 week open labelled, prospective, randomized, multicentric study. The patient will receive either tenofovir, telbivudine or the combination of two drugs. After completion of 24 weeks, the non-responders (ie HBV-DNA > 300 copies/ ml) will be switched to combination arm and will continue receiving tenofovir plus telbivudine for 104 weeks.

ELIGIBILITY:
Inclusion Criteria:

* HBeAg negative at screening
* Documented chronic Hepatitis B
* Treatment naive
* Compensated liver disease

Exclusion Criteria:

* Chronic Hepatitis B with Child Pugh B & C
* HBeAg positive
* Decompensated liver disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-06; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Efficacy of combination of telbivudine plus tenofovir vs monotherapy with either drug alone | 6 Months and 2 Years

SECONDARY OUTCOMES:
Percentage change in serum HBV DNA levels | Baseline and 2 Years
Percentage of patients with ALT normalization | Baseline and 2 Years
Percentage of patients with reduction in HBsAg concentration by >50% | Baseline and 2 Years
Percentage of patients with virological breakthrough | 24 weeks
Percentage of patients with primary treatment failure | 12 weeks
Occurrence of adverse events | 2 Years

CONTACTS AND LOCATIONS:
Overall Officials: Dr S. K. Sarin, MD, DM, Principal Investigator — Institute of Liver & Biliary Sciences
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, India